CLINICAL TRIAL: NCT01129986
Title: A Post Marketing Clinical Study Utilizing DermaStream and Saline for Safety and Efficacy in Venous Stasis Ulcers of the Lower Extremity
Brief Title: A Post Marketing Clinical Study Utilizing DermaStream and Saline in Venous Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EnzySurge (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENZ-DER-003-US
Record Dates: First submitted 2010-05-10; First posted 2010-05-25 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2011-06

CONDITIONS: Venous Stasis Ulcers
Keywords: venous ulcer Dermastream
MeSH Terms: conditions — Varicose Ulcer

ARMS (1):
- Dermastream (Experimental)
  Interventions: Device: DermaStream

INTERVENTIONS:
Device: DermaStream — Five treatment days. On each day DermaStream application for up to 4 hours of saline streaming.

SUMMARY:
An open-label, prospective, controlled, two-step approach, post-marketing clinical study, applying DermaStream with saline streaming, in conjunction with a sustained multi-compression wrap, on healthy individuals and on patients with a venous stasis ulcer of the lower extremity.

ELIGIBILITY:
Inclusion Criteria:

Group A:

* Must be male or female ≥18 years of age.
* Must be a healthy individual with intact skin

Group B:

* Must be male or female ≥18 years of age
* Must have a venous stasis ulcer between the knee and the ankle (including the lateral and medial malleolus). The ulcer must have the typical appearance of venous leg ulceration and the diagnosis of venous origin.
* Ankle Brachial Pressure Index of >0.8 -<=1.2
* Must have a venous leg ulcer between 3 cm up to 5.6 cm maximum and an ulcer duration of 60 days or greater prior to enrollment in the study

Exclusion Criteria:

Group A and Group B:

* Is unable to manage the self-treatment at home
* Is pregnant or is a nursing mother
* Is a woman of child bearing potential who is not using an adequate form of contraception (or abstinent)
* Is < 18 years of age
* With gross morbid obesity (i.e., a Body Mass Index ≥ 50)
* Has a known allergy to any of the drugs and/or dressings that are part of this protocol
* Has previously participated in this study

Group B:

* Has an ulcer that is deemed by the Investigator to be caused primarily by a medical condition other than venous insufficiency (e.g., diabetes, malignant ulceration [Marjolin's ulcer], vasculitis, etc.)
* Has evidence of current clinical infection although colonization is not an exclusion criterion (see definition section)
* Suffers from diabetes mellitus with HbA1c ≥ 10%
* Suffers from clinically significant arterial disease
* Has evidence of the ulcer and/or infection extending to the underlying muscle, tendon, or bone
* Has used any investigational drug(s)/device(s) within 30 days preceding screening or the physician or subject anticipates use of any of these treatments during the 2 weeks following start of the treatment portion of the study
* Has used or is anticipated to use any of the prohibited concomitant medications and treatments, as specified in study protocol, section 9.1.
* Suffers from a condition, other than venous insufficiency or venous hypertension which, in the opinion of the Investigator, would compromise the safety of the subject and/or the quality of the data.
* Suffers from a condition, other than venous insufficiency or venous hypertension which, in the opinion of the Investigator, would seriously interfere negatively with the normal wound healing process.
* Has laboratory values at screening outside ± 20% of the institution's normal range for any parameter other than HbA1c
* If laboratory values are outside ± 20% but the investigator deems the subject acceptable for enrollment, the Principal Investigator may approve the inclusion of the subject as long as there is no evidence of any comorbid condition where comorbidity could influence the trialIs using any of the prohibited concomitant medications or treatments.
* Wound surrounding skin not intact or has signs of active dermatitis or infection
* Wound over-bleeds
* Wound is severely ischemic
* Wound is larger than device aperture diameter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Effect of DermaStream application | Up to 21 days
  Reduction of slough tissue.
Adverse Events | Up to 21 days
  Incidence of investigational product related adverse events
Effect of DermaStream application | Up to 21 days
  Increase of granulation tissue
Effect of DermaStream application | Up to 21 days
  Pain recording on 1-10 scale

SECONDARY OUTCOMES:
Usability | 1-5 days
  Device malfunction reports and device replacements as measures of usability
Wound size | Up to 21 days
  Decrease in wound size at 2 weeks following last treatment day
Quality of Life | Up to 21 days
  Improved "Quality of Life" at 2 weeks following last treatment day

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ihnat, Principal Investigator — S.A.L.S.A, Tucson Arizona
Locations (1):
- S.A.L.S.A, Tucson, Arizona, United States